CLINICAL TRIAL: NCT07050199
Title: Risk Factors Affecting Morbidity and Mortality in Perforated Peptic Ulcer
Brief Title: Risk Factors Affecting Mortality in Perforated Peptic Ulcer
Status: Completed | Type: Observational
Sponsor: Maharajgunj Medical Campus (Other)
Responsible Party: Principal Investigator, Prajjwol Luitel, Co-investigator, Maharajgunj Medical Campus
Other Study IDs: PG-NMC/528/078-079
Record Dates: First submitted 2025-06-14; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Peptic Ulcers
MeSH Terms: conditions — Peptic Ulcer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with peptic ulcer perforation of age > 15 years and <75 years
  Interventions: Procedure: Emergency laparotomy

INTERVENTIONS:
Procedure: Emergency laparotomy — Emergency laparotomy

SUMMARY:
Perforation is one of the most severe and life-threatening complications of peptic ulcer disease. This study aims to evaluate the risk factors associated with postoperative morbidity and mortality in patients undergoing surgery for peptic ulcer perforation, with a focus on the timing of presentation, demographic variables, surgical delay, and their association with postoperative outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with peptic ulcer perforation aged> 15 years and <75 years.
* Patients with duodenal or gastric perforation of peptic ulcer origin.
* Patients who underwent simple closure with omental patch as a standard operative procedure.

Exclusion Criteria:

* Patients treated with conservative management.
* Patients with perforation of peptic ulcer origin at the jejunum, ileum adjacent to Meckel's diverticulum.
* Patients presenting with recurrent perforation or stomal ulcer perforation.

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing emergency laparotomy for peptic ulcer perforation with Graham's patch repair
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Postoperative Morbidity Rate | 12 months (from patient enrollment to completion of follow-up)
  Incidence of postoperative complications (e.g., wound infection, sepsis, anastomotic leak, pneumonia) in patients undergoing surgery for perforated peptic ulcer.
Postoperative Mortality Rate | 12 months (from patient enrollment to completion of follow-up)
  Incidence of death following surgical intervention for perforated peptic ulcer.

CONTACTS AND LOCATIONS:
Locations (1):
- National Medical College and Teaching Hospital, Birgunj, Nepal

IPD SHARING:
Plan to Share IPD: No